CLINICAL TRIAL: NCT01701414
Title: Ultrasound-guided Femoral Nerve Blocks in Elderly Patients With Hip Fractures: a Randomized Controlled Clinical Study
Brief Title: Ultrasound-guided Femoral Nerve Blocks in Elderly Patients With Hip Fractures
Acronym: FNB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210423
Record Dates: First submitted 2012-09-27; First posted 2012-10-05 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2008-02

CONDITIONS: Femoral Neck Fractures; Hip Fractures
Keywords: Femur; Hip; Fracture; Femoral neck; Femoral head
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures; Fractures, Bone | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (SC) (Sham Comparator): The SC group will receive a sham injection of normal saline in order to blind both the participants and the treating physicians. A 7.5-MHz linear transducer will be placed on the side of the affected hip 1cm below the inguinal ligament. 1cm lateral to the ultrasound probe, a 27 gauge needle and syringe will be used to inject 3cc of 0.9% subcutaneously. The SC group will then be cared for by the Emergency Department physicians according to their regular clinical practice.
  Interventions: Drug: Placebo: 3cc of 0.9% Normal Saline
- Femoral Nerve Block (FNB) (Experimental): Participants randomized to the second group, FNB group, will receive an Ultrasound (US) guided femoral nerve block using a Sonosite TitanTM (Sonosite, Inc., Bothell, WA) with a 7.5-MHz linear array transducer. Using this technique, 25ml of 0.5% bupivacaine will be injected along the nerve sheath. The femoral, obturator, and lateral cutaneous nerve are anesthetized with this technique (thus the name "3-in-1 femoral block" is often used), providing maximum analgesia to the hip.
  Interventions: Drug: Femoral nerve block: 25 mL of 0.5% bupivacaine

INTERVENTIONS:
Drug: Femoral nerve block: 25 mL of 0.5% bupivacaine — 25ml of 0.5% bupivacaine will be injected along the nerve sheath. The nerve block will be administered by one of the physician co- investigators all of whom are emergency physicians and all of whom have been trained in the use of ultrasound and ultrasound guided nerve blocks.
  Arms: Femoral Nerve Block (FNB)
Drug: Placebo: 3cc of 0.9% Normal Saline — 1cm lateral to the ultrasound probe, a 27 gauge needle and syringe will be used to inject 3cc of 0.9% NS subcutaneously. The SC group will then be cared for by the Emergency Department physicians according to their regular clinical practice
  Arms: Standard Care (SC)

SUMMARY:
The purpose of this study is to determine if ultrasound guided femoral nerve blocks (localized anesthesia in the upper thigh) provide effective pain relief in adult patients with hip fractures in the emergency department and to determine if femoral nerve blocks can then be used to reduce the use of injected analgesia (anesthesia), therefore also causing fewer adverse effects associated with injected analgesia (such as bruising at the site of injection).

100 patients with hip fractures will be enrolled in the study. Patients will be randomly assigned to receive a femoral nerve block (FNB) plus injected analgesia or standard care (SC), which is injected analgesia alone.

Using guidance from an ultrasound machine, the FNB group will have 20ml of 0.5% bupivacaine (a local anesthetic of long duration) injected into the front of the thigh, at the site of pain. Patients randomized to the SC group will receive an injection of saline (saltwater) so that no neither the patient or the treating physician knows to which group the patient was randomized. All blocks will be performed in the emergency department by an emergency physician trained in the use of ultrasound and ultrasound guided nerve blocks.

Subjects will be asked to rate their pain on a numeric pain scale both before and after intervention (30 min, 60 min, 12 hrs and 24 hrs after injection, as long as the patient is in the ER still). Additional data to be collected includes demographics, vital signs, and course of treatment resulting from the ED visit.

Hypothesis: US-guided femoral nerve blocks can provide effective pain control and possibly decrease or eliminate the need for narcotics.

DETAILED DESCRIPTION:
Hip fractures are a significant cause of morbidity and mortality in the elderly. In the acute setting, safe and effective pain control is of the utmost importance. At present, this is typically achieved with the use of parenteral opioids. However in older individuals, who often have other medical comorbidities, the use of narcotics for pain control must be balanced with their potentially deleterious consequences: namely respiratory depression, hypotension, and mental confusion. Both poor pain control and the use of opioid medications have been associated with acute confusional states in the elderly. 1,2 Regional anesthesia can possibly provide adjunctive or even alternative pain control that is both safe and effective.Femoral nerve blocks, using local anesthetics, have been described as a method to reduce pain and the requirement for systemic analgesia, specifically opioids. Prior research has demonstrated feasibility and effective pain control of the femoral nerve block in the ED setting. Bedside ultrasound (US) can be used to precisely visualize the femoral neurovascular anatomy when performing a femoral nerve block and has distinct advantages when performing this procedure in the ED setting.

Study Objectives The primary aim of this study is to determine the relative effectiveness of ultrasound guided femoral nerve blocks in older adult patients with hip fractures in the emergency department as compared with parenteral narcotics alone. A secondary aim of this study is to determine if femoral nerve blocks reduce both the use of parenteral narcotics and the incidence adverse effects associated with parenteral analgesia (delirium, hypotension, respiratory depression) in hip fracture patients both in the emergency department and during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adults over age 55
* Able to understand and give informed consent
* Comfortable with the experimental protocol as outlined to them by the RA or physician investigator
* Have radiologically confirmed hip fractures: femoral head, femoral neck intertrochanteric, or subtrochanteric femur fractures

Exclusion Criteria:

* Femoral artery grafts on the same side as the fracture
* Extensive lower extremity trauma
* Concurrent tibia-fibula fractures
* Hypersensitivity to local anesthetics or morphine
* Neurovascular injury

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Otto Liebmann, MD, Principal Investigator — Rhode Island Hospital; Francesca Beaudoin, MD, MS, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult ER patients at Rhode Island Hospital were recruited during the course of their clinical care between January 2010 and January 2012.
Pre-assignment Details: Patients were approached after being triaged into the ER system and arrival in a private room but before receiving pain medication for hip fracture. Patients who declined did so because their pain was not severe enough, or they chose not to participate or could not consent, or they were sensitive to morphine (a required component of the study).
Groups:
- Femoral Nerve Block (FNB): Participants randomized to the second group, FNB group, will receive an Ultrasound (US) guided femoral nerve block using a Sonosite TitanTM (Sonosite, Inc., Bothell, WA) with a 7.5-MHz linear array transducer. Using this technique, 25ml of 0.5% bupivacaine will be injected along the nerve sheath. The femoral, obturator, and lateral cutaneous nerve are anesthetized with this technique (thus the name "3-in-1 femoral block" is often used), providing maximum analgesia to the hip.
  Femoral nerve block: 25 mL of 0.5% bupivacaine : 25ml of 0.5% bupivacaine will be injected along the nerve sheath. The nerve block will be administered by one of the physician co- investigators all of whom are emergency physicians and all of whom have been trained in the use of ultrasound and ultrasound guided nerve blocks.
- Standard Care (SC): The SC group will receive a sham injection of normal saline in order to blind both the participants and the treating physicians. A 7.5-MHz linear transducer will be placed on the side of the affected hip 1cm below the inguinal ligament. 1cm lateral to the ultrasound probe, a 27 gauge needle and syringe will be used to inject 3cc of 0.9% subcutaneously. The SC group will then be cared for by the Emergency Department physicians according to their regular clinical practice.
  Placebo: 3cc of 0.9% Normal Saline : 1cm lateral to the ultrasound probe, a 27 gauge needle and syringe will be used to inject 3cc of 0.9% NS subcutaneously. The SC group will then be cared for by the Emergency Department physicians according to their regular clinical practice
Period: Overall Study
Arm/Group | Femoral Nerve Block (FNB) | Standard Care (SC)
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: It was determined that a sample size of 17 in each arm would provide 80% power to detect at least a 33% PID. Sample size was inflated by 10% to account for attrition, missing data, and protocol violations, for a total of 19 subjects in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block (FNB) | Standard Care (SC) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One NRS Rating
Description: Participants report their discomfort using a Numerical Rating Scale (NRS). Pain level is reported as 0 (lowest-no pain) to 10 (highest level of pain). Each patient enrolled in the study reported their level of pain at least once during their participation in the study.
Time Frame: 30 minutes after the block is administered then every 60 minutes until discharge. Desired outcome was a low NRS rating.
Measure: Number; unit: Participants
Arm/Group | Femoral Nerve Block (FNB) | Standard Care (SC)
Number analyzed (Participants) | 18 | 18
Participants | 18 | 18

ADVERSE EVENTS:
Arm/Group | Femoral Nerve Block (FNB) | Standard Care (SC)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes